CLINICAL TRIAL: NCT05832268
Title: The Pelvic Floor Future Study
Brief Title: Pelvic Floor Function After Obstetric Injury to the Anal Sphincter
Acronym: PFF
Status: Enrolling by invitation | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sissel Oversand, Principal investigator, Oslo University Hospital
Other Study IDs: 2019/654
Record Dates: First submitted 2023-03-22; First posted 2023-04-27 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Obstetric Anal Sphincter Injury; Anal Incontinence; Urinary Incontinence; Sexual Dysfunction
MeSH Terms: conditions — Encopresis; Urinary Incontinence; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sphincter damage: Women who suffered an injury to anal sphincter after a vaginal delivery and had a subsequent delivery after this injury
  Interventions: Other: Obstetric Anal Sphincter Injury
- Controls: Women who have had a at least two vaginal deliveries without suffering an injury to the anal sphincter
  Interventions: Other: Obstetric Anal Sphincter Injury

INTERVENTIONS:
Other: Obstetric Anal Sphincter Injury — We will investigate if a new vaginal delivery in those with a previous obstetric anal sphincter injury affects the function of anal musculature negatively

SUMMARY:
The goal of this observational study is to learn more about the effect a pregnancy and delivery has on the function of the anal musculature.We will compare women who had a new delivery after suffering a severe tear in the anal musculature in their first pregnancy, with women who had two or more vaginal deliveries, but did not suffer such an injury.

The main questions we want to answer is:

* can the burden of a new pregnancy and delivery weaken the function of the repaired musculature in a way that might cause symptoms of anal incontinence later in life?
* can a tear in the anal musculature increase the risk of developing urinary incontinence and long term sexual dysfunction?
* should we recommend these women to have a caesarian section instead of a new vaginal delivery?

Participants will be asked to complete an electronic questionnaire with information regarding their pregnancies, deliveries and potential symptoms from anal incontinence, urinary incontinence and sexual dysfunction.

Researchers will compare these two groups to find out if a new vaginal delivery has a negative effect on the function of the anal musculature.

ELIGIBILITY:
Inclusion Criteria:

* Sphincter group: Previous obstetric anal sphincter injury during vaginal childbirth in 2002-2018 and having a subsequent vaginal delivery without such injury
* control group: Two or more vaginal deliveries without obstetric anal sphincter injury

Exclusion Criteria:

* under 18 years
* consent incompetency
* Obstetric anal sphincter injury in subsequent pregnancies
* caesarian section in subsequent pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Study population will be women who had two or more vaginal deliveries at Oslo Universitetssykehus in the time period 2002-2018.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The long-term impact of a new vaginal delivery on anal sphincter function in women with previous obstetric anal sphincter injury. | 5- 20 years
  Number of participants with previous OASI who had a new vaginal delivery will be compared to participants with similar parity, without previous OASI. Differences in anal incontinence symptom score and quality of life will be measured by study questionnaires (St. Marks score, PFDI-20 and PFIQ-7).

SECONDARY OUTCOMES:
Prevalence of urinary incontinence among women with previous OASI compared to women with similar parity without obstetric anal sphincter injury | 5-20 years
  Number of participants who report complaints about urinary incontinence, measured by study questionnaires (PFIQ-7, NFIR, PFDI-20).
The risk of long- term dyspareunia and sexual dysfunction after previous obstetric anal sphincter injury compared to women with similar parity without obstetric anal sphincter injury. | 5-20 years
  Number of participants who report complaints about sexual dysfunction, the degree and type og dysfunction will be measured by study questionnaires (PISQ-12)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Kilaas, M.D, Study Director — Oslo University Hospital; Rune Svenningsen, Ph.D, Study Director — Oslo University Hospital; Sissel Oversand, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
The participant data will only be available to the researchers in charge of this project